CLINICAL TRIAL: NCT06919172
Title: iTBS/fMRI Study of Apex Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Derek Nee, Associate Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 0000033961; R01MH121509 (NIH)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: Transcranial Magnetic Stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- MFG-TMS (Experimental): Transcranial magnetic stimulation to the middle frontal gyrus. 600 pulses delivered in 50 Hz bursts every 5 Hz for 2 seconds repeated every 10 seconds at 80% of resting motor threshold.
  Interventions: Device: transcranial magnetic stimulation
- IPL-TMS (Experimental): Transcranial magnetic stimulation to the inferior parietal lobule. 600 pulses delivered in 50 Hz bursts every 5 Hz for 2 seconds repeated every 10 seconds at 80% of resting motor threshold.
  Interventions: Device: transcranial magnetic stimulation
- S1-TMS (Active Comparator): Transcranial magnetic stimulation to the primary somatosensory cortex. 600 pulses delivered in 50 Hz bursts every 5 Hz for 2 seconds repeated every 10 seconds at 80% of resting motor threshold.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.

SUMMARY:
The objective of this study is to examine the effect of transcranial magnetic stimulation (TMS) on the prefrontal cortex and posterior parietal cortex.

DETAILED DESCRIPTION:
The Comprehensive Control Task (CCT) was designed to examine hierarchical control in a single, well-controlled factorial task. On each trial, participants view a letter surrounded by a colored shape at a particular screen location. Color cues the relevant feature, letter or location, for a block of trials. The first trial of a block requires a decision of whether the stimulus is the first position of a circular sequence (sequence start). Subsequent trials require a decision of whether the viewed stimulus follows the previous stimulus in a circular sequence (sequence 1-back). The letter sequence (T-A-B-L-E-T) and spatial sequence (Top-Bottom Right-Left-Right-Bottom Left-Top) are difficulty-matched.

Shape cues the task to perform. Squares indicate the standard baseline task, and each block begins and ends with baseline trials. Different shapes indicate sub-tasks. In Switching blocks, shape-switches (e.g. from square to circle or circle to square) cue the sequence start task. Shape-repeats cue the sequence 1-back task. In Planning blocks, triangle shapes indicate that the stimulus can be ignored (automatic "no" response). All the while, the last square-shaped stimulus must be retained as a reference for the next square-shaped stimulus. Finally, in Dual blocks, diamond shapes indicate switching (sequence start) and also planning. The reversion back to square shapes requires sequence matching to the distal, previous square.

The design is factorial with stimulus-domain x contextual control x temporal control orthogonally manipulated. Full details of the CCT have been previously described in published work.

The focus in this study will be comparison of MFG-TMS, IPL-TMS, and S1-TMS in an interleaved fMRI-TMS-fMRI design. The logic is to test the apical status of the MFG/IPL through the extent to which TMS impacts other PFC/PPC areas and behavior.

Each experiment will begin with 1 session of the CCT with fMRI to localize TMS targets. Each participant will then perform 3 counter-balanced sessions wherein a different site will be targeted by TMS followed immediately by fMRI on the CCT.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 30
* Right-handed
* Native English speaker or fluent by the age of 6

Exclusion Criteria:

* History of psychiatric disorders
* History of neurological disorders
* Receiving medications for psychiatric or neurological disorders
* Familial history of epilepsy
* Taking any drugs or medications that are pro-epileptic
* Tinnitus
* Women who are pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in PFC-PPC activation | baseline, pre-intervention and immediately after intervention
  blood oxygenation level dependent (BOLD) signal in areas of the prefrontal and posterior parietal cortex assessed with functional magnetic resonance imaging (fMRI) [note, this measure has no units]
Change in PFC-PPC effective connectivity | baseline, pre-intervention and immediately after intervention
  effective connectivity among areas of the prefrontal and posterior parietal cortex in the blood oxygenation level dependent (BOLD) signal assessed with functional magnetic resonance imaging (fMRI) [note, this measure has no units]

SECONDARY OUTCOMES:
Change in contextual control speed | baseline, pre-intervention and immediately after intervention
  behavioral performance (reaction time in milliseconds) on conditions involving contextual control in the comprehensive control task
Change in contextual control accuracy | baseline, pre-intervention and immediately after intervention
  behavioral performance (reaction time in milliseconds) on conditions involving contextual control in the comprehensive control task
Change in temporal control speed | baseline, pre-intervention and immediately after intervention
  behavioral performance (reaction time in milliseconds) on conditions involving temporal control in the comprehensive control task
Change in temporal control accuracy | baseline, pre-intervention and immediately after intervention
  behavioral performance (percent correct) on conditions involving temporal control in the comprehensive control task

CONTACTS AND LOCATIONS:
Overall Officials: Derek Nee, PhD, Principal Investigator — Florida State University
Locations (2):
- United States (2):
  - Florida State University Psychology Department Building, Tallahassee, Florida
  - FSU MRI Facility, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: Yes
Behavioral and imaging data will be shared
Supporting Information: Analytic Code
Time Frame: Within a year following publication of findings
Access Criteria: Behavioral and imaging data will be accessible from NIMH Data Archive
URL: https://nda.nih.gov/edit_collection.html?id=3448